CLINICAL TRIAL: NCT03076671
Title: More Than a Movement Disorder: Applying Palliative Care to Parkinson's Disease
Acronym: MTMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-1400; R01NR016037-01A1 (NIH)
Record Dates: First submitted 2017-02-07; First posted 2017-03-10 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Parkinson Disease; Parkinsonism; Lewy Body Disease; Supranuclear Palsy, Progressive; Parkinsonism Vascular; Multiple System Atrophy; Corticobasal Degeneration; Alzheimer Disease; Frontotemporal Dementia; Primary Progressive Aphasia; Vascular Dementia
Keywords: Palliative Care; Supportive Care; Movement Disorders; Brain Disease; Neurodegeneration; Parkinson's Disease; Alzheimer's Disease
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Lewy Body Disease; Supranuclear Palsy, Progressive; Multiple System Atrophy; Corticobasal Degeneration; Alzheimer Disease; Frontotemporal Dementia; Aphasia, Primary Progressive; Dementia, Vascular; Movement Disorders; Brain Diseases; Nerve Degeneration | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: This is a stepped-wedge design, meaning that during the first year all patients enrolled will continue to receive usual care provided by their neurologist, who is also enrolled in the study. During years 2 and 3, every 6 months, 4-5 neurologists will receive training in supportive and palliative care. The timing of the training will be randomly assigned. Once their neurologist has received training, all of their enrolled patients will be switched to the intervention arm, and be eligible for additional care via telemedicine with the university supportive and palliative care team. During the final year of the study, all the neurologists will have received care, and all of their patients will be in the intervention arm.
  On a separate level, we will be evaluating the effects of training on the enrolled neurologists through assessments of palliative skills, knowledge, and attitudes before and after the training, as well as through qualitative interviews.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (No Intervention): Patients to get usual care from their established neurology care team that is enrolled in the study.
- Standard of Care plus Palliative Care (Experimental): Patients to get usual care, augmented by palliative care, provided by their established neurology care team that is affiliated with the study, with additional support provided by the University of Colorado Denver Neurology Palliative Care team.
  Interventions: Behavioral: Palliative Care
- Clinicians (Experimental): Clinicians enrolled in the study will receive an 8-hour supportive and palliative care training, followed by monthly coaching and the availability of telemedicine visits for enrolled patients with the university neuro-palliative care team. The unit of randomization is the time when they receive training. Four to five clinical practices will receive training every 6 months during years 2 and 3, at which time all of their enrolled patients will be switched from usual care to the intervention arm.
  Interventions: Behavioral: Palliative Care

INTERVENTIONS:
Behavioral: Palliative Care — Palliative care training for community neurologists and use of telemedicine for team-based support of patients
  Other Names: Supportive Care
  Arms: Clinicians; Standard of Care plus Palliative Care

SUMMARY:
This is a two-center (University of Colorado, University of California San Francisco) community-based comparative effectiveness study of outpatient palliative care for Parkinson's disease (PD) and related disorders (progressive supranuclear palsy (PSP), corticobasal degeneration (CBD), multiple systems atrophy (MSA), Lewy Body Dementia (LBD). In September 2018, the study was amended to also include Alzheimer's disease (AD) and related disorders (Frontotemporal Dementia (FTD), Primary Progressive Aphasia (PPA), Vascular Dementia). It will utilize a randomized stepped-wedge design to compare patient and caregiver outcomes between usual care in the community versus usual care augmented by palliative training and telemedicine support to provide other resources (e.g. social work).

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common neurodegenerative illness affecting approximately 1.5 million Americans and is the 14th leading cause of death in the United States. PD is traditionally described as a movement disorder with characteristic motor symptoms (e.g. tremor). However, more recent research demonstrates the impact of nonmotor symptoms such as pain, depression, and dementia on mortality, quality of life (QOL), nursing home placement and caregiver distress. Regarding models of care for PD, evidence suggests that care including a neurologist results in lower mortality and nursing home placement than care solely from a primary care physician. Unfortunately, there is also significant evidence that many of the needs most important to PD patients and their caregivers (e.g. depression, planning for the future) are poorly addressed under current models of care. Palliative care is an approach to caring for individuals with life-threatening illnesses that focuses on addressing potential causes of suffering including physical and psychiatric symptoms, psychosocial issues and spiritual needs. While developed for cancer patients, palliative care approaches have been successfully applied in other chronic progressive illnesses including heart failure and pulmonary disease. To date there have been minimal attempts to apply these principles to PD although evidence suggests that PD patients' unmet needs under current models of care may be amenable to palliative care. A small but growing cadre of centers offer outpatient palliative care for PD with early evidence of efficacy and a randomized trial of an academic-based outpatient palliative care is underway led by investigators on this proposal. While this work is critical to forwarding this field, further work is needed to provide a model that can be widely disseminated. The current proposal addresses this gap by assessing the effectiveness and feasibility of a novel community-based intervention that empowers community neurology practices to improve care for PD patients and caregivers through palliative care training, coaching and telemedicine resources. The investigators hypothesize that this intervention will improve patient QOL and caregiver burden and will prove feasible and acceptable to community providers. The investigators Specific Aims are to: 1) Determine the a) effectiveness and b) feasibility of a novel community-based outpatient palliative care intervention for PD.; 2) Describe the effects of a this intervention on patient and caregiver costs and service utilization; and 3) Identify opportunities to optimize community-based palliative care for this population by: a) describing patient and caregiver characteristics associated with intervention benefits; and b) through direct patient, caregiver and provider interviews. Innovations of the investigators approach include a novel model of providing disease-specific community-based palliative care not dependent on limited palliative specialist resources, a stepped-wedge trial design and use of telemedicine resources to provide multidisciplinary care. The research is significant because it will create a foundation for future community-based dissemination studies in PD and the broader field of palliative care.

In September 2018, supplemental support from NIH was granted in order to explore outcomes among an Alzheimer's dementia population. Alzheimer's disease (AD) is the most common neurodegenerative illness affecting 10% of adults over age 65. This incurable and relentlessly progressive disease affects approximately 1.5 million Americans and is the 6th leading cause of death in the United States. Care for community-dwelling patients with AD is typically focused on the assessment and pharmacologic management of cognitive and behavioral symptoms, although there is growing recognition of the need to expand care to address other issues, including advance care planning. There is significant evidence that many of the most important needs of the AD patients and their caregivers are poorly addressed under current models of care, including management of medical and psychiatric symptoms (e.g. pain and depression), caregiver support, advance care planning, and spiritual wellbeing. Importantly, while the top goal of care for the majority of patients is avoidance of institutionalization, our current models of care invest more resources in institutionalized patients rather than proactively supporting community-dwelling individuals which may prevent institutionalization and reduce overall healthcare costs. Our supplemental study will thus additionally target this population for a 12-month period.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be fluent English Speakers,
* Must be over age 18,
* They must meet United Kingdom (UK) Brain Bank criteria for probable PD, or
* They must meet standard criteria for

  * progressive supranuclear palsy (PSP),
  * corticobasal degeneration (CBD),
  * multiple systems atrophy (MSA),
  * vascular parkinsonism, or
  * Lewy Body Dementia (LBD)
  * Alzheimer's dementia (AD)
  * Primary progressive aphasia
  * Vascular dementia.
* Patients must be at high risk for poor outcomes as defined by the Brief Needs Assessment Tool (BNAT) which screens for psychosocial issues, symptoms, and caregiver burden.
* Caregivers will be identified by asking the patient: "Could (participant) tell us the one person who helps (participant) the most with (participant's) PD outside of clinic?"
* Caregivers may be self-identified in cases of severe dementia in order to obtain data relevant to this vulnerable and underrepresented group.

Exclusion Criteria:

* Unable or unwilling to commit to study procedures;
* Presence of additional chronic medical illnesses which may require palliative services (e.g. metastatic cancer); or
* Already receiving palliative care or hospice services.
* Not expecting to continue care with enrolled physician for at least 6 months.

The investigators have purposefully kept our inclusion/exclusion criteria broad to allow for greater generalizability of results and to ensure inclusion of potentially underrepresented and understudied subgroups.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 783 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of Life Alzheimer's Disease (QOL-AD) | Up to 48 months
  Measures of Quality of Life
Zarit Burden of Care Instrument (ZBI) | Up to 48 months
  Measures of Care Partner Distress

SECONDARY OUTCOMES:
McGill Quality of Life Questionnaire (MQOL) | Up to 48 months
  Measures of Quality of Life
Hospital Anxiety and Depression Scale (HADS) | Up to 48 months
  Measures of mood
Edmonton Symptom Assessment Scale (ESAS_PD) | Up to 48 months
  Measures of symptom burden
Functional Assessment of Chronic Illness Therapy-Spiritual Wellbeing (FACIT-SP 12 Item) | Up to 48 months
  Measures of spiritual wellbeing
Prolonged Grief Questionnaire (PG-12) | Up to 48 months
  Measures of grief (sense of loss)
Semi-structured Qualitative Interview | At 12 months
  Measures of participant views on the study including their outcomes and the implementation of this model of community-based palliative care.
Montreal Cognitive Assessment (MOCA) | At baseline
  Measures of cognitive function
Healthcare Utilization Form | Up to 48 months
  Measures of type and frequency of healthcare utilized
Palliative Performance Scale | Up to 48 months
  Measures of Disease Severity
Clinical Global Impression of Change | Up to 48 months
  Measures of change in disease burden
Treatment Documentation Form | Up to 48 months
  Measures of treatments used for disease management
Modified Caregiver Strain Index | Up to 48 months
  Measures of care partner distress
Needs at End of Life Screening Tool | Up to 12 months
  Detects and measures needs for end of life
Neuropsychiatric Inventory | Up to 6 months
  Measures dementia-related symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Benzi M Kluger, MD, MS, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kluger BM, Katz M, Galifianakis NB, Pantilat SZ, Hauser JM, Khan R, Friedman C, Vaughan CL, Goto Y, Long SJ, Martin CS, Dini M, McQueen RB, Palmer L, Fairclough D, Seeberger LC, Sillau SH, Kutner JS. Patient and Family Outcomes of Community Neurologist Palliative Education and Telehealth Support in Parkinson Disease. JAMA Neurol. 2024 Jan 1;81(1):39-49. doi: 10.1001/jamaneurol.2023.4260. PMID 37955923
- [Derived] Mahes A, Macchi ZA, Martin CS, Katz M, Galifianakis NB, Pantilat SZ, Kutner JS, Sillau S, Kluger BM. The "Surprise Question" for Prognostication in People With Parkinson's Disease and Related Disorders. J Pain Symptom Manage. 2024 Jan;67(1):e1-e7. doi: 10.1016/j.jpainsymman.2023.10.004. Epub 2023 Oct 13. PMID 37838080
- [Derived] Ayele R, Macchi ZA, Dini M, Bock M, Katz M, Pantilat SZ, Jones J, Kluger BM. Experience of Community Neurologists Providing Care for Patients With Neurodegenerative Illness During the COVID-19 Pandemic. Neurology. 2021 Sep 7;97(10):e988-e995. doi: 10.1212/WNL.0000000000012363. Epub 2021 Jun 14. PMID 34489348
- [Derived] Macchi ZA, Ayele R, Dini M, Lamira J, Katz M, Pantilat SZ, Jones J, Kluger BM. Lessons from the COVID-19 pandemic for improving outpatient neuropalliative care: A qualitative study of patient and caregiver perspectives. Palliat Med. 2021 Jul;35(7):1258-1266. doi: 10.1177/02692163211017383. Epub 2021 May 18. PMID 34006157